CLINICAL TRIAL: NCT02492373
Title: Effect of Topical Corticosteroids on the Incidence of Postinflammatory Hyperpigmentation Following Q-switched Nd:YAG 532 nm Laser for Treatment of Facial Lentigines - A Pilot Study
Brief Title: Topical Corticosteroids on the Incidence of Postinflammatory Hyperpigmentation After QsNdYAG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si 033/2015
Record Dates: First submitted 2015-06-27; First posted 2015-07-08 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Lentigines; Post Inflammatory Hyperpigmentation
Keywords: Post inflammatory hyperpigmentation; topical high potency steroid; Qs NdYAG laser
MeSH Terms: conditions — Lentigo; Hyperpigmentation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laser+steroid 2 days before and after laser (Active Comparator): Before lentigines' treatment with Qs Nd:YAG 532 nm laser, topical 0.05% Clobetasol propionate ointment was applied 2 days on the lesion. Then applied 2 days after the treatment.
  Interventions: Drug: topical 0.05% Clobetasol propionate ointment; Device: Q switched Nd:YAG laser 532 nm
- laser+steroid 2 days after laser (Other): Controlled side. Applied topical 0.05% Clobetasol propionate ointment only 2 days after the laser treatment
  Interventions: Drug: topical 0.05% Clobetasol propionate ointment; Device: Q switched Nd:YAG laser 532 nm

INTERVENTIONS:
Drug: topical 0.05% Clobetasol propionate ointment — Apply only on the treated area twice a day as mentions
Device: Q switched Nd:YAG laser 532 nm — Treatment of facial lentigines. The energy using depends on the endpoint of immediate whitening of the lesions.

SUMMARY:
To investigate the benefit of the application of topical high potency steroid on the incidence of post inflammatory hyperpigmentation after laser treatment.

DETAILED DESCRIPTION:
* The incidence of post inflammatory hyperpigmentation (PIH) after treating lentigines with Q-switched Nd:YAG laser was 78.3%.
* It has been found that the incidence of PIH decreased to 40% after applied topical high potency steroid 2 days after the laser treatment.
* By these anti-inflammatory and anti-PIH effects of the high potency steroid, the investigators aimed that the application of steroid 2 days before and 2 days after the laser treatment would be better reduction in the incidence of PIH after Q-switched Nd:YAG laser.

ELIGIBILITY:
Inclusion Criteria:

* Having multiple lentigines on both sides of the face
* Fitzpatrick skin phototype 3-5

Exclusion Criteria:

* Patients with lesions with any clinical suspicion of being pre-cancerous or skin malignancies of any kind
* Patients who have photosensitive dermatoses
* Pregnancy and lactation woman
* Patients with wound infections (herpes, other) on the day of treatment
* Patients with moderate and severe inflammatory acne, Immunosuppressed patients, history of vitiligo
* Patients with unrealistic concerns/expectations and inability to do the appropriate post-operative care

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The incidence of post inflammatory hyperpigmentation | 2 weeks
  By investigator's observation.

SECONDARY OUTCOMES:
Side effects of topical steroid | Follow-up 2, 3, 4, 8, 12 and 24 weeks after the last treatment
  By investigators' observation of telangiectasia, erythema or atrophy.
The patients satisfaction | Follow-up 4, 8, 12 and 24 weeks after the last treatment
  By using Quartile grading scale of improvement; 0 = not improve, 1= 1-25% improvement, 2 = 26-50% improvement, 3 = 51-75% improvement and 4 = 76-100% improvement

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, M.D., Principal Investigator — Department of Dermatology, Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Jun HJ, Cho SH, Lee JD, Kim HS. A split-face, evaluator-blind randomized study on the early effects of Q-switched Nd:YAG laser plus Er:YAG micropeel (combined therapy) versus Q-switched Nd:YAG alone in light solar lentigines in Asians. Lasers Med Sci. 2014 May;29(3):1153-8. doi: 10.1007/s10103-013-1489-9. Epub 2013 Nov 29. PMID 24292155
- [Result] Ho SG, Yeung CK, Chan NP, Shek SY, Chan HH. A comparison of Q-switched and long-pulsed alexandrite laser for the treatment of freckles and lentigines in oriental patients. Lasers Surg Med. 2011 Feb;43(2):108-13. doi: 10.1002/lsm.21045. PMID 21384391
- [Result] Takiwaki H, Shirai S, Kohno H, Soh H, Arase S. The degrees of UVB-induced erythema and pigmentation correlate linearly and are reduced in a parallel manner by topical anti-inflammatory agents. J Invest Dermatol. 1994 Nov;103(5):642-6. doi: 10.1111/1523-1747.ep12398276. PMID 7963648
- [Result] Cheyasak N, Manuskiatti W, Maneeprasopchoke P, Wanitphakdeedecha R. Topical corticosteroids minimise the risk of postinflammatory hyper-pigmentation after ablative fractional CO2 laser resurfacing in Asians. Acta Derm Venereol. 2015 Feb;95(2):201-5. doi: 10.2340/00015555-1899. PMID 24854088